CLINICAL TRIAL: NCT01893346
Title: A Phase I Study to Assess the Pharmacokinetics, Safety and Tolerability of a Single Dose of Ceftazidime-Avibactam (CAZ-AVI) in Children From 3 Months of Age to <18 Years Who Are Receiving Systemic Antibiotic Therapy for Suspected or Confirmed Infection
Brief Title: Safety and Tolerability of Ceftazidime-Avibactam for Pediatric Patients With Suspected or Confirmed Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4280C00014
Record Dates: First submitted 2013-06-26; First posted 2013-07-09 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Systemic Infections
Keywords: Ceftazidime, Avibactam, Anti-Infectives
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAZ-AVI (Experimental): This arm will include 4 cohorts. Patients will be stratified by age.
  Interventions: Drug: CAZ-AVI

INTERVENTIONS:
Drug: CAZ-AVI — Single IV dose of Ceftazidime and Avibactam. Dosage regimen will vary depending on cohort.

SUMMARY:
To assess the pharmacokinetics, safety and tolerability of a single dose of CAZ-AVI in children from 3 months of age to <18 years.

DETAILED DESCRIPTION:
This is a phase I, open-label, single-dose study. The study aims to characterize the pharmacokinetics of CAZ-AVI and assess its safety and tolerability following a single IV dose given to hospitalized pediatric patients receiving systemic antibiotic therapy for suspected or confirmed infection. This study will include 4 cohorts, each consisting of at least 8 evaluable pediatric patients, aged ≥3 months to <18 years, who are hospitalized with infections.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent will be obtained from parent(s) or other legally acceptable representative(s), and informed assent from patient (if age appropriate) will be obtained
2. Male or female children ages ≥3 months to <18 years.
3. Hospitalized, receiving systemic antibiotic therapy for the treatment of a suspected or confirmed infection, and expected to require hospitalization until after the end of treatment (EOT) evaluations are completed.
4. If female and has reached menarche, or has reached Tanner stage 3 breast development (even if not having reached menarche), the patient is practicing appropriate birth control or is sexually abstinent.
5. Likely to survive the current illness or hospitalization.
6. Sufficient intravascular access (peripheral or central) to receive study drug.

Exclusion Criteria:

1. History of hypersensitivity reactions to carbapenems, cephalosporins, penicillin, other β-lactam antibiotics.
2. If female, currently pregnant or breast feeding or has a positive serum β-human chorionic gonadotropin (β-hCG) pregnancy test.
3. Receipt of a blood or blood component (e.g., red blood cells, fresh frozen plasma, platelets) transfusion during the 24-hour period before enrolment.
4. BMI outside the range (below the 5th percentile or above the 85th percentile) for height, age, and weight except for children <2 years of age.
5. Babies born prior to 37 weeks gestation (cohort 4 only).

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MBBS, MRCP, Study Director — AstraZeneca; John Bradley, MD, Principal Investigator — University of California, San Diego
Locations (10):
- United States (10):
  - Research Site, Little Rock, Arkansas
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Louisville, Kentucky
  - Research Site, Omaha, Nebraska
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Houston, Texas
  - Research Site, Morgantown, West Virginia

REFERENCES:
- [Derived] Franzese RC, McFadyen L, Watson KJ, Riccobene T, Carrothers TJ, Vourvahis M, Chan PLS, Raber S, Bradley JS, Lovern M. Population Pharmacokinetic Modeling and Probability of Pharmacodynamic Target Attainment for Ceftazidime-Avibactam in Pediatric Patients Aged 3 Months and Older. Clin Pharmacol Ther. 2022 Mar;111(3):635-645. doi: 10.1002/cpt.2460. Epub 2021 Nov 22. PMID 34687548
- [Derived] Bradley JS, Armstrong J, Arrieta A, Bishai R, Das S, Delair S, Edeki T, Holmes WC, Li J, Moffett KS, Mukundan D, Perez N, Romero JR, Speicher D, Sullivan JE, Zhou D. Phase I Study Assessing the Pharmacokinetic Profile, Safety, and Tolerability of a Single Dose of Ceftazidime-Avibactam in Hospitalized Pediatric Patients. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6252-9. doi: 10.1128/AAC.00862-16. Print 2016 Oct. PMID 27503642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 26 July 2013 Last patient last visit: 09 October 2014
Pre-assignment Details: Eligibility was determined by investigator, prior to enrollment. Patients were selected on the basis of the age requirements for the appropriate cohort and after obtaining written informed consent from the parent or legal guardian and assent from patients (as appropriate). Screening assessments were completed prior to study drug administration.
Groups:
- Cohort 1: aged ≥12 to <18 years 2000 mg ceftazidime and 500 mg avibactam
- Cohort 2: aged ≥6 to <12 years Weight <40 kg: 50 mg/kg ceftazidime and 12.5 mg/kg avibactam Weight ≥40 kg: 2000 mg ceftazidime and 500 mg avibactam
- Cohort 3: aged ≥2 to <6 years Normal renal function or mild renal insufficiency: 50 mg/kg ceftazidime and 12.5 mg/kg avibactam.
  Moderate renal insufficiency: 25 mg/kg ceftazidime and 6.25 mg/kg avibactam
- Cohort 4: aged ≥3 months to <2 years Normal renal function or mild renal insufficiency: 50 mg/kg ceftazidime and 12.5 mg/kg avibactam.
  Moderate renal insufficiency: 25 mg/kg ceftazidime and 6.25 mg/kg avibactam
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 11 | 8 | 8 | 8
Patients Who Received Full Infusion | 8 | 8 | 8 | 8
Completed | 8 | 7 | 8 | 8
Not Completed | 3 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are shown for safety analysis set. The safety analysis set included all patients who received any amount of IV study dose of CAZ AVI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.945 (1.5599) | 8.020 (1.4036) | 3.519 (1.0044) | 0.924 (0.5007) | 6.852 (5.5200)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 6 | 3 | 17
  Male | 3 | 5 | 2 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 8 | 7 | 5 | 7 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3 | 6
  White | 6 | 6 | 7 | 5 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters of Avibactam and Ceftazidime for Cohort 1 and 2: AUC
Description: Key PK parameters were prespecified to be calculated for cohorts 1 and 2. For cohorts 3 and 4 (where children were <6 years of age), sparse sampling scheme was used for PK samples to limit the volume of blood required. PK parameters cannot be derived from these sparse PK samples without population PK analysis. Thus the PK is not described here, but will be reported in a separate population PK report.
Time Frame: Day 1
Population: Pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Cohort 1 / Avibactam: aged ≥12 to <18 years
- Cohort 1 / Ceftazidime: aged ≥12 to <18 years / Ceftazidime
- Cohort 2 / Avibactam; Cohort 2 / Ceftazidime: aged ≥6 to <12 years
Arm/Group | Cohort 1 / Avibactam | Cohort 1 / Ceftazidime | Cohort 2 / Avibactam | Cohort 2 / Ceftazidime
Number analyzed (Participants) | 8 | 8 | 8 | 8
h*ng/mL
  AUC(0-8) | 35140 (33.11) | 219100 (29.69) | 33590 (22.15) | 212400 (16.28)
  AUC(0-t) | 36250 (33.70) | 229200 (30.86) | 34380 (23.37) | 217800 (18.36)
  AUC(0-inf) | 36430 (33.61) | 230600 (30.70) | 34820 (22.62) | 221200 (17.38)

2. Primary Outcome: Pharmacokinetic Parameters of Avibactam and Ceftazidime for Cohort 1 and 2: Cmax
Description: Key PK parameters are shown for cohorts 1 and 2. For cohorts 3 and 4 (where children were <6 years of age), sparse sampling scheme was used for PK samples to limit the volume of blood required. PK parameters cannot be derived from these sparse PK samples without population PK analysis. Thus the PK is not described here, but will be reported in a separate population PK report.
Time Frame: Day 1
Population: Pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 / Avibactam | Cohort 1 / Ceftazidime | Cohort 2 / Avibactam | Cohort 2 / Ceftazidime
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 15090 (52.42) | 79750 (41.81) | 14140 (22.96) | 81270 (17.81)

ADVERSE EVENTS:
Time Frame: From start of study dose infusion of CAZ AVI through the follow up period (Day 2 and Day 3)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 4/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=8) | Cohort 3 (N=8) | Cohort 4 (N=8)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other